CLINICAL TRIAL: NCT01341249
Title: Clinical Trial to Compare the Pharmacokinetic Profiles of DW224aa (Aspartate) Tablet and DW224a (Hydrochloride) Capsule After a Single Oral Administration in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetic Profiles of DW224aa and DW224a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Chang-Soo Cho, DONG WHA PHARMACEUTICAL CO., LTD
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SNUCPT11_DW224aa
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DW224aa (Experimental): DW224aa given by oral administration
  Interventions: Drug: Experimental DW224aa
- DW224a (Active Comparator): DW224aa given by oral administration
  Interventions: Drug: Experimental DW224a

INTERVENTIONS:
Drug: Experimental DW224aa — DW224aa tablet, single dose
  Arms: DW224aa
Drug: Experimental DW224a — DW224a capsule, single dose
  Arms: DW224a

SUMMARY:
The purpose of this study is to compare and explore pharmacokinetics of zabofloxacin, the main component of DW224aa(Test drug) and DW224a(Reference drug).

ELIGIBILITY:
Inclusion Criteria:

* a healthy adult male within the range of 20 to 45 years old at the time of screening
* one with weight of more than 55kg, in the range of IBW 20%

  * IBW(kg)={height(cm)-100}*0.9
* one who understood completely about this study after the detailed explanation is given, decided to volunteer and gave written informed consent to participate in study in compliance with the requirement of the entire protocol.

Exclusion Criteria:

* one with clinically significant disease in liver, kidney, nerve system, respiratory system, endocrine system, blood, tumor, urinary system, cardiovascular system, mental disease or with medical history
* one with gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* one who is allergic or has clinically significant allergic history to the quinolone antibiotics, or to other drugs(Aspirin, antibiotics, etc)
* one who shows the following result in clinical laboratory test: AST,ALT>1.25 times of the upper limit of normal range
* one who has confirmed positive at serological tests (HBs antigen, HCV antibody and HIV antibody)
* one who has drug abuse history or positive result at urine screening tests (cannabinoid, opioid, amphetamine, cocaine, barbiturate, benzodiazepine)
* one who has taken any prescribed drugs, herbal agents or crude drugs within 2 weeks before study drug administration, or who has taken any over-the-counter (OTC) drugs or vitamins (Investigators will determine his eligibility by considering the effect of the drug on his safety or pharmacokinetic results in case other inclusion/exclusion criteria is satisfied.)
* one who has participated in other clinical study within 2 months before study drug administration
* one who donated whole blood within 2 months or component blood within 1 month or who are donated within 1 month before the treatment
* one who drank Over 21 units/week of alcohol or subjects who would not be able to stop drinking alcohol during the hospitalization
* one who are Heavy smoker more than 10 cigarettes/day within 3 months prior to screening or subjects who would not be able to stop smoking during the hospitalization
* one who had a beverage containing caffeine, drank alcohol, or smoked within 48hrs before the hospitalization or who had a beverage containing grapefruits during the hospitalization
* one with clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cmax of zabofloxacin in plasma | Up to 48
AUClast of zabofloxacin in plasma | Up to 48

SECONDARY OUTCOMES:
Tmax of zabofloxacin in plasma | Up to 48h
terminal half-life (t1/2) of zabofloxacin in plasma | Up to 48h
CL/F of zabofloxacin in plasma | Up to 48h

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Han H, Kim SE, Shin KH, Lim C, Lim KS, Yu KS, Cho JY. Comparison of pharmacokinetics between new quinolone antibiotics: the zabofloxacin hydrochloride capsule and the zabofloxacin aspartate tablet. Curr Med Res Opin. 2013 Oct;29(10):1349-55. doi: 10.1185/03007995.2013.825591. Epub 2013 Aug 19. PMID 23865727